CLINICAL TRIAL: NCT03253068
Title: A Phase II Study of Pembrolizumab Plus Amurubicin in Patients With Refractory Small-cell Lung Cancer
Brief Title: Pembrolizumab Plus Amurubicin in Patients With Refractory Small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wakayama Medical University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Hiroaki Akamatsu, Assistant Professor, Wakayama Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-3475-IIT-55441
Record Dates: First submitted 2017-08-12; First posted 2017-08-17 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Small Cell Lung Cancer Extensive Stage
MeSH Terms: interventions — pembrolizumab; amrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab plus amurubicin (Experimental): Pembrolizumab 200mg/body plus amurubicin 40mg/m2, intravenous, every 3 weeks
  Interventions: Drug: Pembrolizumab plus amurubicin

INTERVENTIONS:
Drug: Pembrolizumab plus amurubicin — Pembrolizumab 200mg/body plus amurubicin 40mg/m2, intravenous, every 3 weeks
  Other Names: Keytruda, calsed

SUMMARY:
To explore the overall response rate (ORR) per RECIST 1.1 as assessed by investigators in subjects with refractory small cell lung cancer treated with pembrolizumab (Pembro) plus amurubicin (AMR).

DETAILED DESCRIPTION:
Open, uncontrolled, multi-center, phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed diagnosis of SCLC.
2. Confirmed radiological relapse within 90 days from the last day of first-line chemotherapy.
3. Have adequate tumor tissue sample to test PD-L1 immunohistochemistry.
4. Have measurable disease based on RECIST 1.1 as determined by the site.
5. Be ≥20 years of age on day of signing informed consent.
6. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group
7. Have adequate organ function as indicated by the following laboratory values
8. Is expected to live more than 90 days.
9. Be willing and able to provide written informed consent/assent for the trial.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours from registration.
11. Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days (or longer as specified by local institutional guidelines) after the last dose of study medication.
12. Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in Section 5.7.2- Contraception, starting with the first dose of study therapy through 120 days (or longer as specified by local institutional guidelines) after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 30 days from registration.
2. Is receiving systemic steroid therapy ≤ 3 days from registration or receiving any other form of immunosuppressive medication.
3. Has received prior systemic cytotoxic chemotherapy, biological therapy, OR major surgery within 3 weeks of the first dose of trial treatment; received thoracic radiation therapy of > 30 Gy within 6 months from registration.
4. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody.
5. Has symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis.
6. Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
7. Has had an allogeneic tissue/solid organ transplant.
8. History of noninfectious pneumonitis that required steroids or current active pneumonitis, or any evidence of interstitial lung disease by CT scan.
9. Has received or will receive a live vaccine within 30 days from registration.
10. Has an active infection requiring intravenous systemic therapy and oral administration.
11. Has known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
12. Has known active Hepatitis B, or Hepatitis C.
13. Has any history of prior malignancy, with the exception of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.
14. Has Known history of serious allergy.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days (or longer as specified by local institutional guidelines) after the last dose of trial treatment.
18. Hypersensitivity or allergy to pembrolizumab or any of its excipients, and/or to AMR or any of its excipients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-12-28 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Imaging will be performed every 6 weeks through study completion, an average of 6 months
  Overall response rate will be assessed using RECIST ver1.1 by investigators

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Akamatsu, M.D., Principal Investigator — Third Department of Internal Medicine, Wakayama Medical University; Nobuyuki Katakami, M.D., Ph.D., Principal Investigator — Division of Integrated Oncology, Institute of Biomedical Research and Innovation; Kazuhiko Nakagawa, M.D., Ph.D., Principal Investigator — Department of Medical Oncology, Kinki University, Faculty of Medicine
Locations (1):
- Wakayama Medical University, Wakayama, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akamatsu H, Teraoka S, Hayashi H, Fujimoto D, Hayata A, Haratani K, Ozawa Y, Yoshida T, Iwasa T, Shimokawa T, Tomii K, Nakagawa K, Yamamoto N. Pembrolizumab Plus Amrubicin in Patients With Relapsed SCLC: Multi-Institutional, Single-Arm Phase 2 Study. JTO Clin Res Rep. 2021 May 18;2(7):100184. doi: 10.1016/j.jtocrr.2021.100184. eCollection 2021 Jul. PMID 34590034